CLINICAL TRIAL: NCT01985711
Title: Effects of a Web-Based Collaborative Care Management System (WBCCMS) on Psychosocial Outcomes and Biochemical Outcomes Among Patients With Diabetes and Depression
Brief Title: Web-Based Collaborative Care for Patients With Diabetes and Depression
Acronym: WBCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Tao Hong, PHD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: WBCCFPWDAD
Record Dates: First submitted 2013-11-09; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus, Type 2; Depression
Keywords: Motivational Interviewing; Cognitive Behavioral Therapy; Transtheoretical Model of behavior change; Questionnaires; Telemedicine/*methods; Comorbidity; Diabetes; Glucose/metabolism; Hemoglobin A, Glycosylated; Blood Pressure; Cholesterol, LDL/blood; Quality of life; Depressive Disorder/psychology/*therapy; Randomized Controlled Trials
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Diabetes Mellitus; Depressive Disorder | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- web-based,CBT,MI,TTM, outpatient (Experimental): Participants in web-based collaborative care group will receive 24 weekly 40-minute web-based Cognitive Behavioral Therapy (CBT) sessions, undergo structured Transtheoretical Model of Behavior Change or Motivational interviewing to set up proper life-style and healthy behavior to improve their live quality，conducted on the web. Besides, they will receive usual diabetes outpatient care and web-based diabetes care.
  Interventions: Device: web-based collaborative care; Other: wait-list; Behavioral: usual diabetes outpatient care
- waitlist, usual diabetes outpatient (Other): Participants assigned to the wait-list group will be given usual diabetes outpatient service (diabetic medication guidance and appointment to see doctor as routine, without specific anti-depression therapy). After 6 months, they will receive web-based collaborative care for 6 months too.
  Interventions: Device: web-based collaborative care; Other: wait-list; Behavioral: usual diabetes outpatient care

INTERVENTIONS:
Device: web-based collaborative care — Firstly ,24 weekly 40-minute web-based collaborative care plus usual diabetes outpatient care for 6months.
  Secondly, usual diabetes outpatient care for 6 months.
  Other Names: multidisciplinary care
Other: wait-list — Firstly ,usual diabetes outpatient care for 6 months. Secondly,24 weekly 40-minute web-based collaborative care plus usual diabetes outpatient care for 6months.
  Other Names: usual diabetes outpatient care
Behavioral: usual diabetes outpatient care

SUMMARY:
The goal of this proposal is to integrate depression services and diabetes care methods into a web-based collaborative care system so that a single program can assist patients with diabetes and co-morbid depression. The investigators hypothesized that the effect of the intervention program on (a) decreasing depressive symptomatology; (b) improving biomedical outcomes (e.g., blood lipid profiles,blood glucose, glycosylated hemoglobin, and blood pressure). (c) Increasing healthful behavior (medicine compliance, physical activity, diabetic diet);(d)decreasing unhealthful behavior( sedentary activities, smoking, alcohol addiction); (e) improving quality of life.

DETAILED DESCRIPTION:
Recent study shows that the overall prevalence of diabetes was estimated to be 11.6% (95% confidence interval, 11.3%-11.8%) in the Chinese adult population[1]. Depression is a common comorbidities in patients with diabetes with prevalence rates more than 30%[2, 3]. Co-morbid depression portends worse health outcomes (such as glycemic control, medication adherence, quality of life, physical activity, and blood pressure control，diabetic complication) and increases health care costs[4-6]. But the rate of diabetes-depression recognition and treatment is low. Collaborative primary care model, which involves a multidisciplinary health care team guiding patient-centered care , has been tested in the US and showed a significant reduction of depressive symptoms, improved diabetes care and patient-reported outcomes, and saved money. We aim to developing a web-based collaborative care system and compare the effectiveness of this new collaborative care model with usual diabetes outpatient care for patients with type 2 diabetes and depression in China.

The web-based collaborative care system integrates usual management plan of diabetes and established theories for treating depression and diabetes specific behaviors or affective disorders. Diabetes management plan consists of a meal plan, exercise guidance, oral medications or insulin guidance, health education, supervision and regular blood glucose monitoring. Three main established theories of psychology as follows: 1) Cognitive Behavioral Therapy (CBT); 2) Transtheoretical Model（TTM）of Behavior Change[7]; and 3) Motivational interviewing(MI)[8]. Cognitive behavioral therapy helps people learn to change inappropriate or negative thought patterns and behaviors associated with the illness. Web-based CBT is generally viewed as a very effective form of psychotherapy for treating depression[9-12], which is also effective to manage diabetic stress[13]. Transtheoretical Model of Behavior Change and Motivational interviewing are both evidence-based behavior change techniques to improve diabetes and depression associated healthy behavior (such as taking medicine, physical activity, diabetic diet, drug therapy compliance) and to decrease unhealthy behavior(such as sedentary activities, smoking, alcohol addiction).The intervention will be conducted in a safety-net health system primary care setting.

A randomized controlled trial (RCT) will be conducted to evaluate the effectiveness of culturally adapted diabetes and depression collaborative treatment for reducing depressive symptoms, activating diabetes healthy behaviors, decreasing unhealthy behaviors and improving adherence to diabetes self-care regimens in Chinese with depression and diabetes. Participation in this study will last 12 months. All participants will firstly undergo baseline assessments that will include a 40-minute interview about personal health and feelings. Eligible participants will then be assigned randomly to receive either web-based collaborative care or wait-list. Participants in web-based collaborative care group will receive 24 weekly 40-minute web-based Cognitive Behavioral Therapy (CBT) sessions, undergo structured Transtheoretical Model of Behavior Change or Motivational interviewing to set up proper life-style and healthy behavior to improve their live quality，conducted on the web. Besides, they will receive usual diabetes outpatient care and web-based diabetes care. Participants assigned to the wait-list group will be given usual diabetes outpatient service (diabetic medication guidance and appointment to see doctor as routine, without specific anti-depression therapy). After 6 months, they will receive web-based collaborative care for 6 months too. All participants receiving web-based collaborative care management will also receive supportive patient navigation services and maintenance/relapse telephone monitoring, their assistants (family member; online systems nurse, psychiatrists and endocrinologist) monitor and help them change their behaviors. All participants will undergo follow-up on-site interviews about their status at months 3, 6, 9 and12.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Type 2 Diabetes
* 18 years and older
* be able to surf the internet at least once per week
* willing to give informed consent
* Score >=10 on the PHQ-9

Exclusion Criteria:

* inability to give informed consent
* Already receiving antidepressant treatment(medicine,CBT,et.)
* unwillingness or inability to use the web-based Collaborative Care System.
* Severe and/or terminal physical illness
* Pregnant or breastfeeding
* severe psychiatric disorders (psychotic disorder, major depression and so on) or suicidal tendencies
* Likely to have difficulty completing the forms and questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 items (PHQ-9) score | baseline , 3-month, 6-month,9-month, 12-month
  Depressive symptoms were measured using the nine-item Patient Health Questionnaire (PHQ-9).PHQ-9 scored on a range from 0 to 27, where lower scores represent fewer depressive symptoms.A remission of depression symptoms is indicated with a PHQ-9 score <10 for a period of three consecutive months.

SECONDARY OUTCOMES:
Change in biochemical index | Baseline, 3-month, 6-month, 9-month, 12-month
  We will compare changes in hemoglobin A1c, blood glucose,blood lipids, and blood pressure levels between the immediate intervention group and the wait-list control group over time.Improvement is defined as 10% improvement over baseline.
Chang in quality of life (EuroQol-5D)score | baseline, 3-month, 6-month,9-month, 12-month
  The health-related quality of patients' life was rated with use of the quality-of-life EuroQol-5 Dimensions (EQ-5D)index.
Change in Diabetes-specific stress | Baseline, 3-month, 6-month,9-month, 12-month
  Measured by Problem Areas In Diabetes 5-level questionnaire (PAID-5).
Change in Health behaviours | Baseline, 3-month, 6-month, 9-month, 12-month
  We will assess of smoking behaviours,alcohol consumption, physical activity,and medication taking.
Change in general self-efficacy | Baseline, 3-month, 6-month, 9-month, 12-month
  General self-efficacy is measured by a widely used parsimonious ten-item scale called 'General Self-Efficacy Scale(GSES)',which was developed for use in several cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Hong, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281
- [Background] Roy T, Lloyd CE, Parvin M, Mohiuddin KG, Rahman M. Prevalence of co-morbid depression in out-patients with type 2 diabetes mellitus in Bangladesh. BMC Psychiatry. 2012 Aug 22;12:123. doi: 10.1186/1471-244X-12-123. PMID 22909306
- [Background] Mathew CS, Dominic M, Isaac R, Jacob JJ. Prevalence of depression in consecutive patients with type 2 diabetes mellitus of 5-year duration and its impact on glycemic control. Indian J Endocrinol Metab. 2012 Sep;16(5):764-8. doi: 10.4103/2230-8210.100671. PMID 23087861
- [Background] Ciechanowski PS, Katon WJ, Russo JE. Depression and diabetes: impact of depressive symptoms on adherence, function, and costs. Arch Intern Med. 2000 Nov 27;160(21):3278-85. doi: 10.1001/archinte.160.21.3278. PMID 11088090
- [Background] Lustman PJ, Clouse RE. Depression in diabetic patients: the relationship between mood and glycemic control. J Diabetes Complications. 2005 Mar-Apr;19(2):113-22. doi: 10.1016/j.jdiacomp.2004.01.002. PMID 15745842
- [Background] Lin EH, Katon W, Von Korff M, Rutter C, Simon GE, Oliver M, Ciechanowski P, Ludman EJ, Bush T, Young B. Relationship of depression and diabetes self-care, medication adherence, and preventive care. Diabetes Care. 2004 Sep;27(9):2154-60. doi: 10.2337/diacare.27.9.2154. PMID 15333477
- [Background] Prochaska, J.O., Transtheoretical Model of Behavior Change, in Encyclopedia of Behavioral Medicine. 2013, Springer. p. 1997--2000.
- [Background] Rollnick S, Butler CC, Kinnersley P, Gregory J, Mash B. Motivational interviewing. BMJ. 2010 Apr 27;340:c1900. doi: 10.1136/bmj.c1900. No abstract available. PMID 20423957
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Cuijpers P, Berking M, Andersson G, Quigley L, Kleiboer A, Dobson KS. A meta-analysis of cognitive-behavioural therapy for adult depression, alone and in comparison with other treatments. Can J Psychiatry. 2013 Jul;58(7):376-85. doi: 10.1177/070674371305800702. PMID 23870719
- [Background] Kroenke K, Theobald D, Wu J, Norton K, Morrison G, Carpenter J, Tu W. Effect of telecare management on pain and depression in patients with cancer: a randomized trial. JAMA. 2010 Jul 14;304(2):163-71. doi: 10.1001/jama.2010.944. PMID 20628129
- [Background] Fortney JC, Pyne JM, Edlund MJ, Williams DK, Robinson DE, Mittal D, Henderson KL. A randomized trial of telemedicine-based collaborative care for depression. J Gen Intern Med. 2007 Aug;22(8):1086-93. doi: 10.1007/s11606-007-0201-9. Epub 2007 May 10. PMID 17492326
- [Background] van Bastelaar KM, Pouwer F, Cuijpers P, Riper H, Snoek FJ. Web-based depression treatment for type 1 and type 2 diabetic patients: a randomized, controlled trial. Diabetes Care. 2011 Feb;34(2):320-5. doi: 10.2337/dc10-1248. Epub 2011 Jan 7. PMID 21216855